CLINICAL TRIAL: NCT06898788
Title: Probiotic Administration for Adolescent Depression
Acronym: PAD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 24-41760; R61AT012028 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: probiotics; adolescents; gut microbiome; gut microbiota; fMRI; brain MRI; depression; depressive disorders; youth; young adults
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), 2-arm, single-center, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized into either the Visbiome® or placebo groups through computer-generated randomization at their initial baseline visit, with random block sizes ranging from 2 to 4 and stratification by sex.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Visbiome 450 billion CFU (sachet) twice daily
  Interventions: Drug: Visbiome
- Placebo twice daily (Placebo Comparator): Placebo (maltose sachet) twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Visbiome — Visbiome® is an oral multi-strain probiotic which contains 8 strains: Lactobacillus (L.) paracasei, L. planatrum, L. acidophilus, L. helveticus, Bifidobacterium (B.) longum, B. infantis, B. breve, and Streptococcus (S.) thermophilus.
  Participants will be instructed to consume the powder mixed in water.
  Arms: Probiotic
Drug: Placebo — Participants will be instructed to consume the powder mixed in water (same instructions as the probiotic group).
  Arms: Placebo twice daily

SUMMARY:
This double-blind, placebo-controlled clinical trial will examine the effect of probiotic Visbiome on the brain and gut microbiome of individuals 15 to 24 years of age.

DETAILED DESCRIPTION:
This trial will evaluate the effects of Visbiome 450 billion CFU taken orally twice daily on the biological signature of left hippocampal (HP) resting-state functional connectivity (RSFC) and gut microbiome composition in individuals between the ages of 15 and 24 years.This study will assess the safety and tolerability of Visbiome at this dosage.

Participants will be enrolled in the study for a total of eight weeks and randomized to the probiotic or placebo group. Follow-up assessments will take place every two weeks and will be conducted either through Zoom video visits or in person. The primary outcomes of the study include the effects of the intervention on neural connectivity and gut microbiome composition. Neural connectivity will be assessed by measuring the left HP RSFC using functional magnetic resonance imaging (fMRI). Gut microbiome composition will be evaluated by assessing beta diversity through stool samples collected at baseline and post-intervention.

The safety and tolerability of the intervention will be carefully monitored throughout the study. Adverse events will be systematically collected at each visit, graded for severity, and evaluated for their relationship to the probiotic intervention. Tolerability will be assessed using the Generic Assessment of Side Effects - Probiotics (GASE-P). This measure will be administered at baseline and every two weeks throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Female and male participants 15 to 24 years of age
* Fluency in English
* Access to smartphone, tablet, or computer, on which program "Zoom" can be run for remote visits
* Diagnosed with a primary DSM-5 clinical depressive disorder (Major Depressive Disorder, Persistent Depressive Disorder, or Other Specified Depressive Disorder). The DSM-5 clinical depressive disorder will be confirmed by the Schedule for Affective Disorders and Schizophrenia for School-Aged Children-Computerized Version (K-SADS-COMP)47 to participants <18 years and the Structured Clinic Interview for DSM-5 (SCID-V) to participants ≥18 years.
* Participants must be under the care of a primary care clinician and/or mental health professional
* Currently on SSRI for at least 8 weeks
* BDI-II score greater than 13

Exclusion Criteria:

* Current diagnosis of other DSM-5 mental health disorders except for anxiety disorders and ADHD as long as depressive disorder is the primary diagnosis
* Current medically-treated with stimulant medication for ADHD unless subject is on stable dosage of stimulant medication and there are no plans to change the stimulant medication or dosage for at least 8 weeks.
* Current diagnosis of any Axis II personality disorder(s) as assessed by the K-SADS-COMP or SCID-V.
* Oral probiotic use 1 month prior to phone screening
* Oral or IV antibiotic use 1 month prior to phone screening
* Fermented foods (e.g., yogurt, kombucha) 1 month prior to phone screening
* Oral antioxidant or omega 3 supplements <6 weeks prior to phone screening
* Current alcohol intake greater than 2 drinks per week
* Smoking cigarettes (>5 during last 6 months) or tobacco (pipe or hookah #1 time during last month)
* Any plans to make significant change in diet and lifestyle
* Immunocompromised patients
* Allergies to milk, soy, or yeast
* Tanner Stage <3
* Current active suicidal ideation that requires psychiatric hospitalization or suicidal ideation with plan or intent to attempt suicide as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Prior suicide attempt within past 6 months that required hospitalization and/or visit to the Emergency Department
* History of failure to clinically respond to 2 or more adequate trials of 2 different first-line SSRI antidepressant medications
* Any contraindication to MRI (e.g., braces)
* Pregnancy or any plans to become pregnant during the study is an exclusion criterion for entrance into the study. Women of reproductive capability will be asked about pregnancy or plans to become pregnant. Women of reproductive capability will be asked to employ at least one of the following allowable contraception methods until they complete their second MRI: birth control implant, birth control shot, birth control patch, birth control pill, condom, internal condom, birth control sponge, cervical cap, spermicide, fertility awareness (calendar method), outercourse and abstinence.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Left hippocampus-precuneus resting state functional connectivity | Baseline and week 8
  Measured with fMRI.
Beta diversity | Baseline and week 8
  Gut microbiome measurement
Generic Assessment of Side Effects - Probiotics (GASE-P) | Every 2 weeks from baseline to week 8
  Assesses for tolerability, safety, and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Leung, PhD, RN, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The results of this research will be made available via publication in scientific and medical journals as well as through scientific and medical meetings/conferences where our results will be reported. Publication of data will occur during the time course of this project consistent with normal scientific practices and consistent with NIH policies. Although the final dataset will be stripped of identifiers prior to release for sharing, the investigators believe that there remains the possibility of deductive disclosure of subjects with unusual characteristics. The investigators will thus make the data and associated documentation available to users only under a data-sharing agreement that provides for the following: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Ouwehand AC, Invernici MM, Furlaneto FAC, Messora MR. Effectiveness of Multistrain Versus Single-strain Probiotics: Current Status and Recommendations for the Future. J Clin Gastroenterol. 2018 Nov/Dec;52 Suppl 1, Proceedings from the 9th Probiotics, Prebiotics and New Foods, Nutraceuticals and Botanicals for Nutrition & Human and Microbiota Health Meeting, held in Rome, Italy from September 10 to 12, 2017:S35-S40. doi: 10.1097/MCG.0000000000001052. PMID 29734210
- [Background] Liu RT, Walsh RFL, Sheehan AE. Prebiotics and probiotics for depression and anxiety: A systematic review and meta-analysis of controlled clinical trials. Neurosci Biobehav Rev. 2019 Jul;102:13-23. doi: 10.1016/j.neubiorev.2019.03.023. Epub 2019 Apr 17. PMID 31004628